CLINICAL TRIAL: NCT06403215
Title: The Effect of Chewing Gum and Drinking Fennel Tea on Intestinal Motility After Cesarean Section: A Randomised Controlled Trial
Brief Title: Effect of Chewing Gum and Drinking Fennel Tea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Nurdan Demirci, Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018.2018
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Bowel Ileus; Cesarean Section Complications
Keywords: Cesarean; chewing gum; fennel tea; Bowel sounds
MeSH Terms: conditions — Ileus | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chewing gum group (Experimental): Women in this group chewed sugar-free and non-xylite gum for 15 minutes every two hours (2nd, 4th, and 6th) following the cesarean operation. As a result of their meta-analysis study, a study reported that chewing gum for 15 minutes every two hours until oral intake started bowel sounds in a shorter time. Therefore, in the current study, women chewed gum for 15 minutes every two hours, following two hours after the cesarean operation. The bowel sounds of the women were listened to and their flatulation times were recorded before and after gum chewing for 15 minutes every two hours. When women were allowed oral intake, gum-chewing activity was terminated completely. Data for the first time of flatulation and the bowel sounds were collected by verbally asking women, and these data were recorded in the follow-up form.
  Interventions: Other: Chewing gum group
- Fennel tea group (Experimental): Women in this group started oral intake 6 hours after cesarean delivery and were allowed to drink 2 grams of fennel tea in the 6th, 8th, and 10th hours (a total of 6 grams of fennel tea). Fennel seeds (2 grams) were put into 150 ml water, boiled at a temperature of 100 °C, and left for 20 minutes. Women were then instructed to drink the tea. Bowel sounds were recorded every 2 hours, before and after drinking the fennel tea. The time of the first flatulation and the first bowel sounds were determined by asking the women themselves and this information was then recorded using the study form.
  Interventions: Other: Fennel tea group
- Chewing gum+Fennel tea group (Experimental): Women in this group chewed sugar-free and non-xylite gum for 15 minutes every two hours (2nd, 4th, and 6th) following the cesarean operation. As a result of their meta-analysis study, a study reported that chewing gum for 15 minutes every two hours until oral intake started bowel sounds in a shorter time.Women were then instructed to drink the tea. Bowel sounds were recorded every 2 hours, before and after drinking the fennel tea. The time of the first flatulation and the first bowel sounds were determined by asking the women themselves and this information was then recorded using the study form.
  Interventions: Other: Chewing gum+Fennel tea group
- Control group (Experimental): Researcher sounded in bowel movement as hospital protocols.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Chewing gum group — Women in this group chewed sugar-free and non-xylite gum for 15 minutes every two hours (2nd, 4th, and 6th) following the cesarean operation.
  Arms: Chewing gum group
Other: Fennel tea group — Women in this group started oral intake 6 hours after cesarean delivery and were allowed to drink 2 grams of fennel tea in the 6th, 8th, and 10th hours (a total of 6 grams of fennel tea).
  Arms: Fennel tea group
Other: Chewing gum+Fennel tea group — Women in this group both chewed sugar-free and non-xylite gum for 15 minutes every two hours (2nd, 4th, and 6th) following the cesarean operation and started oral intake 6 hours after cesarean delivery and were allowed to drink 2 grams of fennel tea in the 6th, 8th, and 10th hours (a total of 6 grams of fennel tea).
  Arms: Chewing gum+Fennel tea group
Other: Control group — No intervention
  Arms: Control group

SUMMARY:
Aim: Postoperative ileus after cesarean section is a problem that significantly prolongs hospital stay and increases perioperative costs. The ability of postoperative fennel tea consumption to produce bowel movement is unclear and needs to be studied. This study aimed to determine the effect of chewing gum and drinking fennel tea on intestinal motility after cesarean section.

Methods: The study was conducted in postnatal care wards between January 2018 and April 2018. Simple randomization was used to assign women to the study arms. Data were collected during Pregnancy Constipation Diagnostic Scale, Data Collection and Follow-up Form were collected.

DETAILED DESCRIPTION:
Study Sample This parallel, monocenter, randomized controlled experimental study was conducted between January 2018 and April 2018 with the CONSORT guidelines in four maternity units in Türkiye. Inclusion criteria for the study were as follows: Healthy, women who had a cesarean section under general anesthesia, received primary school education at least, did not have a chronic systemic disease, had no problems during pregnancy, had no history of allergy, had a body mass index (BMI) of 18.50-24.99 kg/m2, with no previous abdominal operation, and no complications during the operation.

Participants and Setting After being included in the study, the women were registered as a participant and the study was carried out using opaque sealed envelopes numbered sequentially. The study was carried out with four different groups determined by 22 factorial trial levels. The sample size was determined as a total of 120 participants at 80% power and 95% confidence interval in consideration of the meta-analysis conducted on the data of the subjects. Two different interventions- chewing gum and drinking fennel tea - were conducted in this study.

Intervention Chewing gum group Women in this group chewed sugar-free and non-xylite gum for 15 minutes every two hours (2nd, 4th, and 6th) following the cesarean operation. As a result of their meta-analysis study, a study reported that chewing gum for 15 minutes every two hours until oral intake started bowel sounds in a shorter time. Therefore, in the current study, women chewed gum for 15 minutes every two hours, following two hours after the cesarean operation. The bowel sounds of the women were listened to and their flatulation times were recorded before and after gum chewing for 15 minutes every two hours. When women were allowed oral intake, gum-chewing activity was terminated completely. Data for the first time of flatulation and the bowel sounds were collected by verbally asking women, and these data were recorded in the follow-up form.

Fennel tea group Women in this group started oral intake 6 hours after cesarean delivery and were allowed to drink 2 grams of fennel tea in the 6th, 8th, and 10th hours (a total of 6 grams of fennel tea). Fennel seeds (2 grams) were put into 150 ml water, boiled at a temperature of 100 °C, and left for 20 minutes. Women were then instructed to drink the tea. Bowel sounds were recorded every 2 hours, before and after drinking the fennel tea. The time of the first flatulation and the first bowel sounds were determined by asking the women themselves and this information was then recorded using the study form.

Data collection The amount of fluid taken by the patients was measured with a glass. The amount of urine removed was calculated by checking the patient's bladder. The urinary catheter was removed at the 6th hour.

Ethical Statement The study was conducted in accordance with the Declaration of Helsinki and were approved by Ethics Committees (Protocol No: 09.2017.586). All patients signed informed consents.

Data Analysis Chi-square and Fisher tests were used to compare categorical data. Spearman's rank correlation coefficient was used to analyze and compare the statistical data. A value of p<0.05 was accepted for the statistical significance of the comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Without chronic disease
* women who had a cesarean section under general anesthesia
* received primary school education at least
* women had no problems during pregnancy
* who had no history of allergy
* who had a body mass index (BMI) of 18.50-24.99 kg/m2
* no previous abdominal operation
* no complications during the operation.

Exclusion Criteria:

* age<18 years
* multiparous women
* who had a cesarean section under spinal anesthesia
* spontaneous onset of labor
* who had a chronic systemic disease
* who had problems during pregnancy
* who had any history of allergy
* who had a body mass index (BMI) of <24.99 kg/m2
* who had a previous abdominal operation, and complications during the operation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
bowel sounds | 12 hours
  Bowel sounds were recorded every 2 hours.
flatulation | 24 hours
  .The time of the first flatulation were determined by asking the women themselves and this information was then recorded using the study form.
defecation | 48 hours
  .The time of the first defecation were determined by asking the women themselves and this information was then recorded using the study form.

CONTACTS AND LOCATIONS:
Overall Officials: Rüveyda Ölmez Yalazı, PhDc, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No